CLINICAL TRIAL: NCT05459753
Title: Cholinergic Mechanisms of Attentional-motor Integration and Gait Dysfunction in Parkinson Disease (UDALL)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, Professor of Radiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00197590; 1P50NS123067-01 (NIH)
Record Dates: First submitted 2022-07-01; First posted 2022-07-15 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease; Progressive Supranuclear Palsy
Keywords: Parkinson's Disease; Parkinson; Parkinson's; Freezing of Gait; FOG; PIGD
MeSH Terms: conditions — Parkinson Disease; Supranuclear Palsy, Progressive | interventions — Fluorine-18; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; dihydrotetrabenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson's Disease (Experimental): Individuals with idiopathic Parkinson's disease.
  Interventions: Radiation: (18)F]fluoroethoxybenzovesamicol ([(18)F (FEOBV) PET; Radiation: Dihydrotetrabenazine (DTBZ) PET

INTERVENTIONS:
Radiation: (18)F]fluoroethoxybenzovesamicol ([(18)F (FEOBV) PET — Participants will receive an injection of 8 mCi [18F]FEOBV PET tracer and undergo a CT of the head.
Radiation: Dihydrotetrabenazine (DTBZ) PET — Participants will receive an injection of 15 mCi [11C]DTBZ PET tracer and undergo a CT of the head.

SUMMARY:
To perform a prospective cohort study with [(18)F]fluoroethoxybenzovesamicol (FEOBV) brain PET at baseline and 2-year follow-up in PD subjects at risk of conversion to non-episodic and episodic (falls and FoG) PIGD motor features and cognitive changes at the same time points.

DETAILED DESCRIPTION:
Postural instability and gait difficulty (PIGD) motor and cognitive changer features are common in Parkinson disease (PD), and a significant cause of treatment-refractory disability. Accumulating evidence implicates cholinergic systems dysfunctions as significant contributors to gait and balance and cognitive impairment. During the initial funding period, the investigators established the vesicular acetylcholine transporter (VAChT) ligand FEOBV, which uniquely assesses cholinergic terminal density in high density regions such as the striatum. Recent cross-sectional findings suggest that people with Parkinson's (PwP) participants with isolated falls and those with freezing of gait (FoG) status share common cholinergic deficits in the thalamus (lateral geniculate nucleus (LGN)) and striatum (caudate) with more extensive striatal, limbic, and prefrontal VAChT reductions in PwP with FoG. These data suggest that SChI deficits are a common denominator in the etiology of falls and FoG. These results emphasize the need to understand PIGD, falls, and FoG as products of cholinergic projection dysfunctions within the framework of failing Attentional-Motor Integration (AMI) combined with failures of additional multisensory and cognitive integration.

There is novel preliminary data that cholinergic deficits of the medial geniculate nucleus (MGN) and the entorhinal cortex (ERC) are robustly associated with non-episodic PIGD deficits. These results imply a significant role of impaired sensorimotor integration underlying non-episodic PIGD motor features in PwP. There is also have novel data that cholinergic changes in the cingulo-opercular task control network (COTC) are a robust correlate of cognitive changes in PwP. The overarching goal of this project is to investigate the evolution of cholinergic deficits within multisensory, cognitive and motor integration brain regions and development of PIGD features and cognitive deficits in PwP. This study will perform a prospective cohort study with FEOBV brain PET at baseline and 2-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 for normal control subjects (Male/Female) and ≥45 for Parkinson's disease (PD), Progressive supranuclear palsy (PSP), or Alzheimer's disease (AD) participants (Male/Female).
* For normal control subjects, no significant neurological or psychiatric symptoms and normal neuropsychological examination for age.
* PD diagnosis (with or without Mild Cognitive Impairment/dementia) will follow the Movement Disorder Society-revised clinical diagnostic criteria for PD or Parkinson-PSP patients.
* Modified Hoehn and Yahr stages 1-4.
* AD subjects meeting the criteria listed in Guy M. McKhann et al.
* All PD subjects are required to have nigrostriatal dopaminergic denervation as demonstrated by vesicular monoaminergic transporter type-2 (VMAT) [18F]9-fluoropropyl-(+)-dihydrotetrabenazine (DTBZ) positron emission tomography (PET) imaging. This may be based on a prior DTBZ PET scan or the DTBZ PET scan performed as part of this study.

Exclusion Criteria:

* Disorders which may resemble PD, such as dementia with Lewy bodies, vascular dementia, normal pressure hydrocephalus, multiple system atrophy, corticobasal ganglionic degeneration, or toxic causes of parkinsonism. The use of the Movement Disorder Society-revised clinical diagnostic criteria will mitigate the inclusion of PD subjects with atypical parkinsonism.
* Subjects on neuroleptic, anticholinergic (trihexyphenidyl, benztropine), or cholinesterase inhibitor drugs. Subjects with prior exposure to disallowed medications may be eligible if there has been an interval of > 2 months off these medications.** Note that patients on pimavanserin will be eligible.
* Evidence of a large vessel stroke in a clinically relevant area (cerebral cortex, basal ganglia, thalamus) or mass lesion on structural brain imaging (MRI or CT).**
* Participants in whom MRI is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant.**
* Severe claustrophobia precluding MR or PET imaging.**
* Subjects limited by previous participation in research procedures involving ionizing radiation.**
* Pregnancy (test within 48 hours of each PET session) or breastfeeding.**
* History of deep brain stimulation surgery.**
* Suicidality (responses 2 or 3 for question 9 on the Beck Depression Inventory).
* Subjects from the previous U-M Udall Center cohort who have developed a contraindication for neuroimaging procedures (Exclusion criteria #4 - #9) or have started taking cholinergic medications (Exclusion criterion #3) will be eligible to continue their participation in clinical assessments but will not be referred to neuroimaging assessments.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Interval change on the Unified Parkinson's disease rating scale (UPDRS) motor rating scale over a 2-yr period | At Baseline and at 2-year follow up
  Interval change baseline vs 2-yr follow-up on the UPDRS motor score. UPDRS motor section is scored from 0-132, with higher scores indicating more severe motor symptoms.
Cholinergic brain PET FEOBV PET distribution volume ratio (DVR) interval change over a 2-yr period | At Baseline and at 2-year follow up
  Interval change baseline vs 2-yr follow in cholinergic brain FEOBV PET DVR
Cognitive 2-yr interval change on the Montreal Cognitive Assessment (MoCa) cognitive scale | At Baseline and at 2-year follow up
  Interval change baseline vs 2-yr follow-up on the Montreal Cognitive Assessment (MoCa) cognitive scale. The MoCa is scored out of 30, with higher scores indicating better cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Albin, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan - Michigan Medicine, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Barr J, Vangel R, Kanel P, Roytman S, Pongmala C, Albin RL, Scott PJH, Bohnen NI. Topography of Cholinergic Nerve Terminal Vulnerability and Balance Self-Efficacy in Parkinson's Disease. J Integr Neurosci. 2024 Sep 24;23(9):178. doi: 10.31083/j.jin2309178. PMID 39344233